CLINICAL TRIAL: NCT05404321
Title: Establishment of an ex Vivo Tumor Collection of Triple-negative Breast Cancers in Order to Validate the Interest of Innovative Therapies and the Search for Predictive Biomarkers of Response to Treatment
Acronym: TRIPLEX
Status: Recruiting | Type: Observational
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A02676-35
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Triple Negative Breast Cancer; Organoid
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient with early stage triple negative breast cancer
  Interventions: Other: Establishment of ex vivo breast cancer organoid models

INTERVENTIONS:
Other: Establishment of ex vivo breast cancer organoid models — This study includes 2 steps: The constitution of a collection of tumor and blood samples and the analysis of the ex vivo response of the tumor samples to the treatments for the development of functional tests and the research of predictive biomarkers of this response

SUMMARY:
Initially described in 2009 on LGR5 positive stem cells from intestine, organoids correspond to a 3D cell culture that preserves the organization and part of the initial function of the organ from which the cells were derived. They use the proliferation and differentiation properties of stem cells cultured in a three-dimensional matrix.

These principles have been adapted to many human organs, including the breast. These culture conditions have thus allowed the establishment of cancer organoid lines that have the advantages of rapid amplification, a high rate of establishment success and unlimited proliferation potential. They are transfectable and cryopreservable. They are very close morphologically and genetically to the tumor from which they derive. Very recently, the in vivo response of orthotopic xenograft models of breast cancer organoids has been correlated to the in vitro response of these same organoids. In addition, the in vitro response of various of these models to PARP inhibitors was linked to the presence of the BRCA1/2 mutant signature, highlighting the potential of these models to predict patient response to these treatments.

Furthermore, one study demonstrated the value of using organoids derived from metastatic gastrointestinal tumors to predict patient response to cancer treatments (100% sensitivity, 93% specificity, 88% positive predictive value, and 100% negative predictive value.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patient with early stage (I-III) triple negative breast cancer who needs to have clips placed before neoadjuvant chemotherapy
* Patient affiliated to a social security system
* Proficiency in French language,
* Patient having signed the consent to participate in the study.

Exclusion Criteria:

* Pregnant women
* Persons deprived of liberty or under guardianship (including curatorship)
* History of any other clinically active malignancy in the last 5 years prior to inclusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with early stage (I-III) triple negative breast cancer who needs to have clips placed before neoadjuvant chemotherapy
Sampling Method: Probability Sample
Enrollment: 163 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of establishment of exploitable organoids tumor | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Centre François Baclesse, Caen, France

REFERENCES:
- [Derived] Divoux J, Florent R, Jacobs M, Lequesne J, Grellard JM, San C, Grossi S, Kerdja K, Clarisse B, Boudier G, Cherifi F, Briand M, Dolivet E, Johnson A, Dubois B, Harter V, Lacroix J, Raboutet C, Marie B, Rousseau N, Blanc-Fournier C, Vaur D, Figeac M, Poulain L, Weiswald LB, Emile G. The TRIPLEX study: use of patient-derived tumor organoids as an innovative tool for precision medicine in triple-negative breast cancer. BMC Cancer. 2023 Sep 19;23(1):883. doi: 10.1186/s12885-023-11362-8. PMID 37726786